CLINICAL TRIAL: NCT02445326
Title: A Multi-Center, Randomized, Double-Masked, Vehicle Controlled Phase 3 Study Evaluating the Efficacy and Safety of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model (CAC®)
Brief Title: OTX-14-007: A Phase 3 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-14-007
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Chronic Allergic Conjunctivitis
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Other: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of the signs and symptoms of chronic allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Has a positive history of ocular allergies and a positive skin test reaction to a perennial allergen and a seasonal allergen
* Has a positive bilateral CAC reaction to a perennial allergen within minutes of instillation

Exclusion Criteria:

* History of refractive surgery (including LASIK procedures)
* History of retinal detachment, diabetic retinopathy, or active retinal disease
* Presence of an active ocular infection or positive history of an ocular herpetic infection at any visit
* Use any of the disallowed medications during the period indicated
* History of IOP increase as a result of steroid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Vehicle: PV (placebo drug delivery vehicle)
Period: Overall Study
Arm/Group | OTX-DP | Placebo Vehicle
Started | 35 | 38
Completed | 33 | 37
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP | Placebo Vehicle | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Full Range); unit: years] | 38.2 [19 to 66] | 36.3 [18 to 62] | 37 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 18 | 24 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 10 | 12 | 22
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 4 | 6
Iris Color [Count of Participants; unit: Participants]
  Blue | 4 | 1 | 5
  Brown | 26 | 32 | 58
  Hazel | 1 | 0 | 1
  Green | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 3 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.68 (1.032) | 2.66 (0.861)

2. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.87 (1.040) | 2.74 (0.690)

3. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 7 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.70 (0.938) | 2.74 (0.679)

4. Primary Outcome: Conjunctival Redness Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 7 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.52 (0.641) | 1.80 (0.764)

5. Primary Outcome: Conjunctival Redness Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.48 (0.698) | 1.75 (0.786)

6. Primary Outcome: Conjunctival Redness Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=None
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 35 | 38
units on a scale | 1.44 (0.710) | 1.76 (0.766)

ADVERSE EVENTS:
Arm/Group | OTX-DP | Placebo Vehicle
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 3/35 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (N=35) | Placebo Vehicle (N=38)
Adverse Events (General disorders) | 3 (4) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No